CLINICAL TRIAL: NCT06166589
Title: The Efficacy and Safety of Second-line Zimberelimab and SIRIOX Chemotherapy for Patient With Previously AG Chemotherapy Treated Pancreatic Cancer: A Prospective, Single Arm, Phase II Clinical Study
Brief Title: Second-line Zimberelimab and SIRIOX Chemotherapy for Patient With Previously AG Chemotherapy Treated Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSPAC-04
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Previously AG Chemotherapy Treated Pancreatic Cancer
Keywords: pancreatic cancer; chemotherapy; PD-1 therapy; second-line treatment
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — zimberelimab; Oxaliplatin; S 1 (combination); Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zimberelimab in combination with SIROX chemotherapy (Experimental)
  Interventions: Drug: Zimberelimab; Drug: Oxaliplatin; Drug: S-1; Drug: Irinotecan

INTERVENTIONS:
Drug: Zimberelimab — Zimberelimab, 240mg, day1. Every 3 weeks as a cycle.
Drug: Oxaliplatin — Oxaliplatin 60mg/m2, day1、day8. Every 3 weeks as a cycle.
Drug: S-1 — S-1(BSA < 1.2m2, 40 mg/day; BSA = 1.2~1.4 m2, 60 mg/day; BSA = 1.4~1.6 m2, 80 mg/day; BSA > 1.6 m2, 100 mg/day; bid, day1-14). Every 3 weeks as a cycle.
Drug: Irinotecan — Irinotecan, 130 mg/m2, day 1, day 8. Every 3 weeks as a cycle.

SUMMARY:
This is a prospective, single arm, phase II clinical study investigating second-line Zimberelimab and SIROX chemotherapy for patient with previously AG chemotherapy treated pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients are at least 18 years old when signing the informed consent, both male and female.
* Patients with pancreatic cancer progressing after first-line AG regimen chemotherapy, including patients with advanced pancreatic cancer progressing after first-line AG regimen chemotherapy and patients with recurrence and metastasis after radical pancreatic cancer surgery assisted by AG regimen chemotherapy.
* Having not been previously treated with oxaliplatin, S-1, irinotecan and PD-1/L1 antibody.
* According to the judgment of the attending physician, it is appropriate to receive sepalizumab treatment.
* According to RECIST1.1, Patients must have measurable target lesions examined by CT or MRI.
* ECOG PS score: 0-1.
* Expected survival time ≥3 months.
* All screening period laboratory tests should be performed as required by the protocol and within 14 days prior to the first dose.
* Women of childbearing age must take a serum pregnancy test within 3 days before the first medication, and the result is negative. Female Patients of reproductive age and male Patients whose partners are women of reproductive age must agree to use highly effective methods of contraception during the study period and for 180 days after the last dose of the study drug.
* Voluntarily participate in clinical research and sign informed consent.

Exclusion Criteria:

* Patients have any active autoimmune disease or a history of autoimmune disease (such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism;Patients with vitiligo or complete remission of asthma in childhood without any intervention after adulthood can be included;Patients with asthma requiring medical intervention with bronchodilators cannot be included);
* Patients are using immunosuppressants, or systemic, or absorbable topical hormone therapy for immunosuppression purposes (dose > 10mg/day prednisone or other therapeutic hormones), and continue to use within 2 weeks before enrollment;
* Severe allergic reactions to all drugs and excipients involved in the study;
* Clinical cardiac symptoms or diseases that have not been well controlled, such as: (1) NYHA2 or higher heart failure (2) unstable angina (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* Urine routine suggests proteinuria ≥++, or confirmed 24-hour urinary protein ≥1.0g;
* Patients have active infection or unexplained fever >38.5 degrees during screening and before the first dose; 7. The Patients have congenital or acquired immune deficiency (such as HIV infection), or active hepatitis (hepatitis B reference: HBsAg positive, and HBV DNA detection value exceeds the upper limit of normal value; hepatitis C reference: HCV antibody positive, and HCV virus titer detection value exceeds the upper limit of normal value);
* The Patients have used other drugs in clinical trials within 4 weeks before the first dose;
* The Patients have suffered from other malignant tumors in the past or at the same time;
* The Patients may receive other systemic anti-tumor treatment during the study period;
* The patients with bone metastasis have received palliative radiotherapy in the area >5% of the bone marrow area within 4 weeks before participating in the study;
* The Patients have been vaccinated less than 4 weeks before the study dose or may be vaccinated during the study period;
* In the judgment of the researchers, the Patients have other factors that may lead to the forced termination of the study, such as other serious diseases (including mental diseases) requiring combined treatment, serious laboratory abnormalities, accompanied by family or social factors that may affect the safety of the Patients, or the collection of data and samples. In the judgment of the researchers, there are other factors that may affect the results of the study or lead to the forced termination of the study, such as alcoholism, drug abuse, drug abuse, other serious diseases (including mental illness) that need combined treatment, serious abnormalities in laboratory tests, and family or social factors that may affect the safety of medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | one year
  Objective response rate based on RECIST v1.1

SECONDARY OUTCOMES:
adverse events | two years
  adverse events evaluation based on NCI-CTCAE 5.0
DCR | one year
  Disease control rate evaluation based on RECIST v1.1
PFS | two years
  Progression free survival time
OS | three years
  overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Liang Liu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.